CLINICAL TRIAL: NCT06653075
Title: Role of Clinical Overjet for Mandibular Advancement: a Prospective Study
Brief Title: Mandibular Advancement Planning Based on Clinical Overjet
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Giorgio Gastaldi, Associate Professor, IRCCS Ospedale San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OJ2024
Record Dates: First submitted 2024-10-17; First posted 2024-10-22 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Overjet; Class II Division 1 Malocclusion
MeSH Terms: conditions — Overbite; Malocclusion, Angle Class II | interventions — Mandibular Advancement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional anchorage (Active Comparator): Skeletal class II patients treated by Herbst Appliance with traditional dental anchorage
  Interventions: Procedure: mandibular advancement with acrylic splint Herbst Appliance
- skeletal anchorage (Experimental): Skeletal class II patients treated by Herbst Appliance with skeletal anchorage
  Interventions: Procedure: mandibular advancement with acrylic splint Herbst Appliance

INTERVENTIONS:
Procedure: mandibular advancement with acrylic splint Herbst Appliance — Mandibular advancement with acrylic splint Herbst Appliance

SUMMARY:
This Prospective study aims to simulate the maximum mandibular advancement in class II patients treated by Herbst MTH Appliance on the base on clinical overjet.

Initial intraoral scans will be uploaded in Suresmile software, the upper incisors will be virtually aligned and the mandible will be advancement until an anterior occlusal contact will be reached. This virtual advancement will be compared to the real advancement obtained at the end of the Herbst phase.

This protocol will be applied to two groups: one with traditional dental occlusion, the second one with Skeletal anchorage reinforcement and elastic chains

ELIGIBILITY:
Inclusion Criteria:

* ANB>=4°
* Overjet >=4 mm
* Class II malocclusion ( bilateral class II molar relation, at least half a cusp)

Exclusion Criteria:

* tooth agenesis
* poor oral hygiene
* previous orthodontic treatments
* systemic disease or bone pathology

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Planned mandibular advancement (mm) | 1 year
  The "planned mandibular advancement" will be evaluated on the STL of the arches by simulating a sagittal mandibular advancement , until an anterior occlusal contact will be reached

SECONDARY OUTCOMES:
Obtained mandibular advancement (mm) | 1 year
  The obtained mandibular advancement will be evaluated comparing the Sagittal position of the Pogonion (according to cephalometric pancherz's analysis) on the lateral ceph before and after the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Vita-Salute San Raffaele University, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Manni A, Lupini D, Cozzani M. Les elastiques intermaxillaires a ancrage osseux dans une malocclusion de Classe II asymetrique : une etude de cas. Int Orthod. 2017 Jun;15(2):263-277. doi: 10.1016/j.ortho.2017.03.012. Epub 2017 Apr 25. No abstract available. French. PMID 28389184
- [Result] Manni A, Boggio A, Gastaldi G, Cozzani M. Is significant mandibular advancement possible after the peak of puberty? Dento-osseous palatal expansion and the STM4 technique (Skeletal Therapy Manni Telescopic Herbst 4 miniscrews): A case report. Int Orthod. 2024 Jun;22(2):100868. doi: 10.1016/j.ortho.2024.100868. Epub 2024 Mar 11. PMID 38471383
- [Result] Manni A, Boggio A, Caldara G, Gastaldi G, Cozzani M. Herbst appliance with four-miniscrew anchorage for mandibular advancement after the pubertal peak. J Clin Orthod. 2024 Aug;58(8):505-513. No abstract available. PMID 39307830
- [Result] Manni A, Pasini M, Mauro C. Comparison between Herbst appliances with or without miniscrew anchorage. Dent Res J (Isfahan). 2012 Dec;9(Suppl 2):S216-21. doi: 10.4103/1735-3327.109762. PMID 23814587
- [Result] Manni A, Mutinelli S, Cerruto C, Cozzani M. Influence of incisor position control on the mandibular response in growing patients with skeletal Class II malocclusion. Am J Orthod Dentofacial Orthop. 2021 May;159(5):594-603. doi: 10.1016/j.ajodo.2020.02.014. Epub 2021 Feb 7. PMID 33563504
- [Result] Manni A, Migliorati M, Calzolari C, Silvestrini-Biavati A. Herbst appliance anchored to miniscrews in the upper and lower arches vs standard Herbst: A pilot study. Am J Orthod Dentofacial Orthop. 2019 Nov;156(5):617-625. doi: 10.1016/j.ajodo.2018.11.015. PMID 31677670